CLINICAL TRIAL: NCT05092191
Title: Efficacy of Cannabinoids to the Current Standard Treatments on Symptom Relief in Persons With Multiple Sclerosis: Randomized Controlled Trial
Brief Title: Cannabis as a Complementary Treatment in Multiple Sclerosis
Acronym: CANSEP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Multiple Sclerosis Society of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-9017; 431518 (Other Grant/Funding Number: Canadian Institutes of Health Research); AA1 (Other Grant/Funding Number: Multiple Sclerosis Society of Canada)
Record Dates: First submitted 2021-09-01; First posted 2021-10-25 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Randomized Controlled Trials as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CBD alone (Experimental): * Dosage form : Softgel
  * Dosage & frequency : 40 mg /day of CBD up to 200 mg in two doses a day
  * Duration : 4 weeks of treatment followed by 12 additional weeks of follow up.
  Interventions: Drug: Cannabis oil vs placebo
- THC alone (Experimental): * Dosage form : Softgel
  * Dosage & frequency : 4 mg /day of THC up to 20 mg in two doses a day
  * Duration : 4 weeks of treatment followed by 12 additional weeks of follow up.
  Interventions: Drug: Cannabis oil vs placebo
- THC and CBD combined (Experimental): * Dosage form : Softgel
  * Dosage & frequency : 40 mg /day of CBD up to 200 mg and 4 mg /day of THC up to 20 mg in two doses a day
  * Duration : 4 weeks of treatment followed by 12 additional weeks of follow up.
  Interventions: Drug: Cannabis oil vs placebo
- Placebo (Placebo Comparator): * Dosage form : Softgel
  * Dosage & frequency : caps of placebo twice a day
  * Duration : 4 weeks of treatment followed by 12 additional weeks of follow up.
  Interventions: Drug: Cannabis oil vs placebo

INTERVENTIONS:
Drug: Cannabis oil vs placebo — Eligibility, Screening and Baseline (T0):
  Candidates will be seen by both research staff and a neurologist. Full written informed consent will be obtained before completing questionnaires and administering physical and medical evaluations. If eligibility is confirmed, a blood sample will be collected followed by participant randomisation .
  Follow-up visits:
  Randomized participants come back after 4 weeks (T1) for the same assessments administered at T0. Only participants who had a decrease in their level of spasticity can continue their participation in the same allocated arm for an additional period of 12 weeks.
  At the end of the additional period of 12 weeks (T2), another visit is scheduled for a last assessments which are the same as T0 and T1.
  Throughout study, courtesy calls will be scheduled and standard care for MS will also be offered to ensure participants 'safety and well-being.
  Other Names: Randomized Controlled Trial

SUMMARY:
Multiple sclerosis (MS) is an inflammatory disease of the central nervous system (CNS) afflicting over 77,000 Canadians. Unfortunately, the therapeutic arsenal to relieve MS symptoms is limited. It is therefore essential to develop better approaches to treat the symptoms of MS. The use of cannabis for recreational purposes is now legal in Canada. However, for many years, people with Multiple Sclerosis (PwMS) have used cannabis either to relax, to reduce pain and spasticity, or to improve sleep and daily functioning. Currently, there is little scientifically established evidence that cannabis works on these symptoms in people with MS. It is therefore important to carry out studies to better understand the efficacy Δ-9-tetrahydrocannabinol (THC), and cannabidiol (CBD) on MS symptoms . THC is known for its analgesic, neuroprotective and anti-inflammatory properties and CBD seems to have positive effects on anxiety and cognitive abilities (memory, concentration).

For this study, investigators hypothesize that administering different doses of THC alone, CBD alone, and THC and CBD combined will result in a significant beneficial effect on spasticity relief compared to placebo.

DETAILED DESCRIPTION:
The aim of this study is to document,

1. The efficacy of THC and CBD, alone and in combination, as add-on therapies to the current standard treatments for relief of spasticity and other symptoms in PwMS (muscle spasms and stiffness);
2. Assess the tolerability profile of THC and CBD, alone and in combination, when used in PwMS;
3. Identify the mechanisms underlying such therapeutic and adverse effects of different types of cannabis-based medicines in PwMS,

Participants will initially receive THC 4mg/day or CBD 40mg/day or THC/CBD combination (THC 4mg and CBD 40mg/day), or placebo, on the first day. Dose will be increased up to 20mg (THC) and 200mg (CBD) per day, if well tolerated. Participants will receive the allocated treatment for a total of 4 weeks, followed by an additional 12 weeks of treatment for responders who will be identified as patients who had a decrease from baseline in spasticity of at least one point on the Numerical Rating Scale . THC and CBD will be taken as oil softgels in two divided doses per day. Cannabis extract and placebo will taste and look exactly the same.

To protect from all contingencies and to minimize the risk of adverse reactions, the presence of adverse events will be evaluated at each research visit, as well as through courtesy calls between visits. If any mental or physical symptoms occur that require medical attention, the PwMS will be referred as required to an attending neurologist, psychiatrist, or other specialists .

ELIGIBILITY:
Inclusion Criteria:

Participants must meet the following criteria:

1. Diagnosed with MS (any subtype), for at least six months, by a MS neurologist, according to the recent version of the McDonald criteria;
2. Spasticity due to MS of at least one-month duration and not relieved with current therapy, at a level of 4 or more on the numerical rating scale (NRS);
3. Stable dose of standard therapies for at least 30 days prior to the screening visit and willingness for these to be maintained for the duration of the study;
4. Aged 21 years or older;
5. Ability (in the investigator's opinion) and willingness to comply with all study requirements;
6. Ability to speak and read French or English (grade-nine level of language required);

Exclusion Criteria:

Participants will be excluded if any of the following criteria are met:

1. Concomitant disease with symptoms of spasticity, or that may have influenced their level;
2. Received a botulinum toxin injection within four months prior to the screening visit or unwillingness to stop receiving botulinum toxin injections for the duration of the study;
3. Use of cannabis or cannabinoid-based medications within 7 days of study entry and unwillingness to abstain for the duration of the study;
4. History of schizophrenia, other psychotic illness or other significant psychiatric disorder other than anxiety or depression associated with their underlying condition;
5. Alcohol or substance use disorder other than nicotine;
6. History of epilepsy or recurrent seizures;
7. Hypersensitivity to cannabinoids or any of the excipients of the study medication;
8. Clinically relevant cardiac dysfunction within the last 12 months or had a cardiac disorder that, in the opinion of the investigator would put the subject at risk of a clinically relevant arrhythmia or myocardial infarction;
9. Impaired renal function i.e., serum creatinine clearance lower than 50 ml/min;
10. Significantly impaired hepatic function, at visit 1, in the investigator's opinion and/or had liver function tests of equal to or greater than three times the upper limit of normal;
11. Pregnancy or breastfeeding;
12. Men with history of fertility problems and who plan to conceive at any time in the future;
13. Any participant who plans to conceive either at screening or while enrolled in the study;
14. Inability (or unwillingness) of women of childbearing potential and men to use a medically acceptable form of contraception throughout the study duration;
15. Inability to use a medically acceptable form of contraception throughout the study duration; m) any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, may influence the result of the study, or the subject's ability to participate in the study;
16. Intention to travel internationally, or to donate blood during the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Spasticity patient reported change assessment | Change from Baseline Patient reported spasticity at 28 weeks and 16 weeks
  Patient-reported spasticity: a Numerical rating scale - 0 (No pain) to 10 (worst pain)

OTHER OUTCOMES:
Spasticity change Clinician assessment | Change from Baseline Clinician evaluation spasticity at 28 weeks and 16 weeks
  Spasticity: Ashworth scale -1 (normal) to 4 (rigid)
Pain change assessment | Change from Baseline pain at 28 weeks and 16 weeks
  Pain: Pain Effects-1 (Not at all) to 4 (extreme)
Mobility Change assessement | Change from Baseline mobility at 28 weeks and 16 weeks
  Mobility: Timed 25-Foot Walk test
Fatigue change assessement | Change from Baseline fatigue at 28 weeks and 16 weeks
  Fatigue: Modified Fatigue Impact Scale-0 (never) to 4 (always)
Sleep change assessement | Change from Baseline sleep at 28 weeks and 16 weeks
  Sleep: Pittsburgh Study Quality sleep Index-0 (no difficult) to 3 (severe)
Drowsiness change assessement | Change from Baseline Drowsiness at 28 weeks and 16 weeks
  Drowsiness: Epworth Sleepiness scale-0 (no chance) to 3 (High chance)
Bowel /Bladder dysfunction change assessement | Change from Baseline Bowel/Bladder dysfunction at 28 weeks and 16 weeks
  Bowel /Bladder dysfunction: Bowel/Bladder Control Scale-0 (not at all) to 4 (Daily)
Sexual dysfunction change assessement | Change from Baseline Sexual dysfunction at 28 weeks and 16 weeks
  Sexual dysfunction: Sexual Satisfaction Scale-0 (Extremely Satisfied) to 6 (Extremely Dissatisfied)
Restless Legs Syndrome change assessement | Change from Baseline Restless Legs Syndrome at 28 weeks and 16 weeks
  Restless Legs Syndrome - 4 (V.severe) to 0 (None)
Mental Health disorder change assessement | Change from Baseline Mental Health at 28 weeks and 16 weeks
  Mental Health issues: Mental Health inventory-1 (All of the time) to 6 (None of the time)
Anxiety/Depression change assessement | Change from Baseline Anxiety/Depression at 28 weeks and 16 weeks
  Anxiety/Depression: Hospital Anxiety and Depression-0 to 3 (highest level)
Cannabis use disorder assesssment | Cannabis use disorder : assessment at only baseline
  Cannabis use disorder : diagnosis
Cognition change assessement | Change from Baseline cognition at 28 weeks and 16 weeks
  Cognition tests
Quality of life change assessement | Change from Baseline Quality of life at 28 weeks and 16 weeks
  Quality of life: Health Status Questionnaire (Higher scores indicate better health)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Duquette, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- CRCHUM, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Zertal A, Alami Marrouni K, Arbour N, Jutras-Aswad D, Pomey MP, Rouleau I, Prat A, Larochelle C, Beaulieu P, Chamelian L, Sylvestre MP, Morin D, Ouellette JS, Frejeau N, Duquette P. Efficacy of cannabinoids compared to the current standard treatments on symptom relief in persons with multiple sclerosis (CANSEP trial): study protocol for a randomized clinical trial. Front Neurol. 2024 Jul 24;15:1440678. doi: 10.3389/fneur.2024.1440678. eCollection 2024. PMID 39114536